CLINICAL TRIAL: NCT05373030
Title: Immunogenicity and Safety of a Recombinant Adenovirus Type-5-vectored COVID-19 Vaccine in Healthy Adults (18-80 Years Old) Finished 3 Doses Inactivated COVID-19 Vaccine: a Randomised, Double-blind, Parallel Controlled, Clinic Trial
Brief Title: Sequential Immunization With Recombinant Adenovirus Type-5-vectored COVID-19 Vaccine in Health Adults Based on 3 Doses Inactivated COVID-19 Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS-NCOVIM-ZJ001
Record Dates: First submitted 2022-05-12; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Immunogenicity and Safety of a Recombinant Adenovirus Type-5-vectored COVID-19 Vaccine Using for Sequential Immunization

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant adenovirus type-5-vectored COVID-19 vaccine (Experimental)
  Interventions: Biological: Recombinant adenovirus type-5-vectored COVID-19 vaccine
- Inactivated COVID-19 vaccine (Active Comparator)
  Interventions: Biological: Recombinant adenovirus type-5-vectored COVID-19 vaccine

INTERVENTIONS:
Biological: Recombinant adenovirus type-5-vectored COVID-19 vaccine — One dose COVID-19 vaccine

SUMMARY:
COVID-19 is a novel coronavirus infection caused by respiratory droplets and contact transmission. With the spread of the epidemic, it has become a serious threat to global public health. China has launched a full range of vaccination including the third dose of homologous and sequential booster immunization. To further improve COVID-19 vaccine immunization strategy, we start the clinic research about sequential Immunization With Recombinant Adenovirus Type-5-vectored COVID-19 Vaccine in Health Adults Based on 3 Doses Inactivated COVID-19 Vaccine in Zhejiang province.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers aged 18 and above at the time of screening;
2. Obtain the informed consent of the volunteers and sign the informed consent;
3. Volunteers are able and willing to comply with the requirements of the clinical trial protocol and complete the 6-month study follow-up;
4. Have received 3 doses of Sinovac/Beijing Biological Novel Coronavirus inactivated vaccine with an interval of 6-9 months.

Exclusion Criteria:

1. Patients with history or family history of convulsion, epilepsy, encephalopathy and mental illness;
2. Those who are allergic to any of the components of the study vaccine, have had a severe allergic reaction to the vaccine in the past, a history of allergy or asthma;
3. Serious adverse events related to vaccination occurred after previous vaccination; 4) Positive urine pregnancy test in women during lactation or childbearing age;

5) Acute febrile disease, infectious disease, SARS history; 6) Axillary body temperature > 37.0℃; 7) Suffering from serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension and uncontrolled medication (systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥110mmHg when measured on site); 8) Patients with serious chronic diseases that are in the advanced stage and cannot be controlled smoothly, such as diabetes and thyroid diseases; 9) Congenital or acquired angioedema/neuroedema; 10) Urticaria 1 year before receiving the test vaccine; 11) No spleen or functional no spleen; 12) Patients with chronic obstructive pulmonary disease, pulmonary fibrosis and other pulmonary abnormalities; 13) History of novel coronavirus infection/illness; 14) Have traveled to medium or high risk areas or left the country in the past 21 days; have a history of novel Coronavirus 2019-epidemiological contact; 15) The researcher made a judgment based on various medical, psychological, social or other conditions that might be contrary to the test protocol or affect the subjects to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-14 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reactions (AR) in 0-14 days after immunization | 14 days
  Incidence of adverse reactions (AR)
Geometric mean titer (GMT) of neutralizing antibody against SARS-COV-2 at 14 days after immunization | 14 days
  Geometric mean titer (GMT) of neutralizing antibody against SARS-COV-2

CONTACTS AND LOCATIONS:
Locations (1):
- Xihu District Center for Disease Control and Prevention, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Zhang H, Xu N, Xu Y, Qin P, Dai R, Xu B, Wang S, Ding L, Fu J, Zhang S, Hua Q, Liao Y, Yang J, Hu X, Jiang J, Lv H. Safety and immunogenicity of Ad5-nCoV immunization after three-dose priming with inactivated SARS-CoV-2 vaccine in Chinese adults. Nat Commun. 2023 Aug 8;14(1):4757. doi: 10.1038/s41467-023-40489-2. PMID 37553338